CLINICAL TRIAL: NCT01923584
Title: A Phase 2A Trial of EPI-743 for Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIPD
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPI-743 400mg (Active Comparator): EPI-743 at a dose of 400 mg three times daily
  Interventions: Drug: EPI-743 400mg
- EPI-743 200mg (Active Comparator): EPI-743 at a dose of 200 mg three times daily
  Interventions: Drug: EPI-743 200mg

INTERVENTIONS:
Drug: EPI-743 400mg
  Arms: EPI-743 400mg
Drug: EPI-743 200mg
  Arms: EPI-743 200mg

SUMMARY:
The purpose of this study is to evaluate the effects of EPI-743 in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Age 40 - 75
3. Ambulatory with or without assistance
4. Hoehn and Yahr Scale score of 1 - 3
5. Patient able to consent and comply with protocol requirements
6. Abstention from use of Coenzyme Q10, vitamin E, Azilect and Idebenone two weeks prior to enrollment and during course of treatment with EPI-743

Exclusion Criteria:

1. Allergy to EPI-743 or sesame oil
2. Allergy to vitamin E
3. Clinical history of bleeding or abnormal baseline PT/PTT
4. Diagnosis of any other neurologic disease
5. Malignancy within past two years
6. Pregnant or plans to become pregnant
7. Concomitant ophthalmologic disease
8. History of stroke
9. History of brain surgery
10. Inability to undergo MRI scan or MRS
11. Hepatic insufficiency with LFTs greater than two times upper limit of normal
12. Renal insufficiency requiring dialysis
13. End stage cardiac failure
14. Fat malabsorption syndromes precluding drug absorption
15. Use of anticoagulant medications, azilect

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Visual function | 3 months
  electroretinogram and color vision

SECONDARY OUTCOMES:
Neurologic function | 3 months
  UPDRS subscales
Motor function | 3 months
  UPDRS subscales
Brain metabolites | 3 months
  Magnetic Resonance spectroscopy (MRS)
Cognitive function | 3 months
  Montreal Cognitive Assessment (MoCA)
Mood | 3 months
  Beck Depression Inventory (BDI)
Disease biomarkers | 3 months
  Blood biomarker levels
Safety | 3 months
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States